CLINICAL TRIAL: NCT00172133
Title: An 18-Month Open Label Extension Study (OLES) of the Safety and Efficacy of Recombinant Human Parathyroid Hormone, rhPTH(1-84), ALX1-11, in Women With Postmenopausal Osteoporosis Who Participated in Protocol ALX1-11-93001 (TOP Study)
Brief Title: Open Label Extension Study of PREOS
Acronym: OLES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-11-002
Expanded Access: Available
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Osteoporosis
Keywords: Post-menopausal; Osteoporosis; Parathyroid Hormone; PTH; ALX1-11
MeSH Terms: conditions — Osteoporosis | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All patients entering the study will receive 100mcg daily for up to 6 months, making their total exposure 24 months
  Interventions: Drug: ALX1-11 (drug)

INTERVENTIONS:
Drug: ALX1-11 (drug) — 100 mcg PTH(1-84) injected subcutaneously daily in either the thrigh and abdomen.
  Other Names: PREOS

SUMMARY:
This is an Open Label Extension Study (OLES) for patients who participated in the 18 month double-blind, placebo-controlled, Phase III trial (Protocol ALX1 11 93001 the TOP Study) studying the effect of ALX1-11, recombinant human parathyroid hormone, rhPTH(1-84), on vertebral fracture incidence. The primary objective of this study is to evaluate the safety of continued dosing with ALX1-11, up to a maximum of 24 months, in postmenopausal osteoporotic women who participated in Protocol ALX1 11 93001.

DETAILED DESCRIPTION:
Effects of ALX1-11 on bone mineral density (BMD) have been documented in a dose-finding Phase II clinical trial in osteoporotic postmenopausal women, supplemented with calcium and Vitamin D3 but without any other treatment for osteoporosis. The anabolic effects of ALX1-11 in the lumbar vertebrae were statistically significant after the 12-month treatment period and more pronounced than any approved therapy. Additionally, animal studies have shown that the new bone formed by treatment with ALX1 11 is of good quality both histologically and biomechanically.

The primary objective of this OLES is to evaluate the safety of continued dosing with ALX1-11, up to a maximum of 24 months, in postmenopausal osteoporotic women who participated in Protocol ALX1-11-93001. A secondary objective is to assess the change in vertebral BMD and compare the changes observed in patients who received ALX1-11 or placebo in Protocol ALX1-11-93001.

Patients will receive 100 µg/day of ALX1-11 daily via subcutaneous injection in this study. Patients should continue the study drug dosing frequency they were following at the end of Protocol ALX1-11-93001.

To enhance their safety, all patients will continue to take their daily supplements of 700 mg calcium and 400 IU Vitamin D3 prior to and during this OLES. Patients whose calcium supplement was discontinued during Protocol ALX1-11-93001 should maintain that discontinuation during this OLES. However upon completion of ALX1-11 dosing in the OLES, oral calcium supplement at a dose of 700 mg each morning should be restarted and maintained for the remainder of the OLES. Additional supplemental calcium and/or Vitamin D3 will not be permitted. A daily multivitamin supplement may be taken during the study. However, the multivitamin must contain no more than 200 mg/day calcium and 400 IU/day Vitamin D3. Patients will be monitored for the development of hypercalcemia and/or hypercalciuria and managed as described in Appendices 4 and 5.

There will be a stopping rule in this OLES. Any patient who reaches a BMD T score of -0.5 or above, at the site or sites (vertebral, total hip, or femoral neck) that were used in the qualification of the patient for Protocol ALX1 11-93001, will stop ALX1-11 treatment. The patient must continue on calcium and Vitamin D3 and be followed for the remainder of this 18-month OLES. At the time of discontinuation, the patient must complete the Month 18 evaluations (Appendix 1A or 1B).

The Clinical Advisory Board (CAB) used in Protocol ALX1-11-93001 will be involved in reviewing any patient issues that arise in this OLES. This group will provide not only continuity of care for all the patients, but also enhanced and consistent safety monitoring for patients participating in the OLES.

ELIGIBILITY:
Inclusion Criteria:

* Women who completed 18 months of treatment in Protocol ALX1-11-93001; or
* Women prematurely discontinued from Protocol ALX1-11-93001 who want to participate in OLES for the events listed below must have their clinical course reviewed and approved by the CAB for enrollment into the OLES:

  * Clinical or incident lumbar vertebral fractures as assessed by the central imaging organization
  * Clinical or incident hip fracture
  * Confirmed bone loss at A/P lumbar vertebra or total hip or femoral neck as assessed by the central imaging organization
* Body weight below 40 kg
* Development of an exclusion criterion in Protocol ALX1-11-93001
* It must be accepted by patients whose clinical courses are reviewed by the CAB that participation in OLES may require additional tests at baseline and/or during the study to ensure their utmost safety.
* Women with the ability to self-administer a daily injection or have a designee who will give the injections;
* Women who are capable of understanding and giving written, voluntary informed consent before the start of open-label dosing with ALX1-11.

Exclusion Criteria:

A. History or Concurrent Illness:

Disorders of Immunity Endocrine system Gastrointestinal system Kidney and collecting system Liver, biliary tract and pancreatic systems Musculoskeletal system

* Patients with chronic, active joint disease requiring more than one intra-articular injection every 6 months Neoplasia
* Patients who have had squamous or basal cell carcinoma of the skin may enter this study if:

  1. The lesion(s) were fully resected with clear margins described in a written report by a pathologist, and
  2. The patient has had no recurrence of lesions for at least one year from the time of the original resection.

     Nervous system Vascular, respiratory and cardiac system *Significant diseases or disorders are determined by history, physical exam or laboratory tests and judged by the Principal Investigator to be significant.

     B. Concurrent Medication:

     Patients may not use any of the following therapies while they are enrolled in this OLES without permission from the Sponsor and the PMO:
     * Tetracycline antibiotics for four weeks prior to bone biopsy
     * Any PTH analogs [e.g., rhPTH(1-84), PTH(1-34), PTHrP and analogs]
     * Fluoride
     * Strontium
     * Phenytoin for seizure control
     * Any investigational drug other than ALX1-11
     * Anabolic steroids or androgens
     * Active Vitamin D3 metabolites and analogs, e.g., calcitriol
     * Systemic corticosteroids, more than 5 mg/day prednisone or a systemic corticosteroid formulation equivalent to 5 mg/day prednisone

  1. A patient who has been enrolled into the OLES and needs to receive an acute bolus of steroids (oral or injectable) for a self-limited illness may continue treatment in the study if the following requirements are met:
  1. Exposure to steroids will be limited to no more than 30 consecutive days
  2. The maximal dose of steroid (prednisone equivalent) must be limited to no more than 225 mg (7.5 mg each day for 30 days)
  3. The illness is acute in nature and is not expected to recur during the remaining period of the study

     * Bisphosphonates, including investigational bisphosphonates
     * Calcitonin
     * Estrogen replacement therapy by oral, transdermal or intramuscular administration
     * SERM drugs, e.g., tamoxifen, raloxifene, Evista
     * Vaginal application of estrogen-containing creams unless the dose is:

       1. conjugated estrogen or estradiol: maximum of 0.5 g twice each week (total of 1.0 g weekly)
       2. Estrace (Ogen): maximum of 1.0 g twice each week (total of 2.0 g weekly)
     * Daily inhaled corticosteroid unless dose is equivalent to <1200 µg/day of beclomethasone
     * Cytostatics, e.g., azathioprine, recombinant human tumor necrosis fusion (Fc) protein, monoclonal antibody against tumor necrosis factor (e.g., remicade [infliximab]
     * Methotrexate

       1. The antimetabolite, methotrexate, which interferes with DNA synthesis, repair and cellular replication should not be used by patients participating in this OLES.
     * In general, immunomodulatory agents with antiproliferative activity are not permitted as a concomitant medication in this OLES.
     * Intra-articular injections

       1. Patients may receive a maximum of one intra-articular injection (ONE JOINT ONLY) every 6 months while participating in this OLES. The joint that is injected may be a different joint every 6 months. The dose of corticosteroid injected should not exceed the anti-inflammatory equivalent dose of Prednisone 40 mg suspension. The dose and volume should be adjusted downward as appropriate to the size of the joint.
     * Provera is an acceptable concomitant medication when used according to the label instructions

     Patients may be enrolled in this OLES if they have been stabilized on the following therapy for the specified amount of time:
     * Thyroid Hormone (<0.1 mg/day thyroxine) therapy for at least 6 months If taking > 0.1 mg/day but < 0.2 mg/day, must have serum TSH level 1. > 0.1mU/L. Patients will be excluded if they are taking doses of > 0.2 mg/day.

       2. However, if a patient has had a minimal change in L-thyroxine dose of < 0.025 mg/day within 6 months of the baseline visit, and has been on this new dose for at least 2 months, the patient may be enrolled in this study. The patient's history with L-thyroxine must be clearly documented in the source documents.

       3. If a patient requires an increase in their thyroid replacement dose, as recommended by a physician who is caring for the patient, after enrollment in this OLES, the patient must have a TSH and T4 level within 3 months of the dose change to ensure the patient does not become hyperthyroid
     * Stable dosage of thiazide for at least 3 consecutive months

     C. Laboratory Values and Physical Examination Findings:

     - Serum calcium greater than 10.7 mg/dL (2.66 mmol/L) at baseline will be managed as outlined in Appendix 4

     - Urinary calcium to creatinine ratio greater than or equal to 1 at baseline will be managed as outlined in Appendix 5
     * Elevated total serum alkaline phosphates (> 400 U/L) at baseline will be managed as outlined in Appendix 6 except as noted for Latin and South American countries.
     * Any other clinically significant abnormal value as judged by the investigator

     D. Substance Abuse:

     Alcohol and/or drug abuse

     E. Compliance:

     Suspected or confirmed poor compliance in completing clinical trial evaluations and/or clinical trial required questionnaires

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1683 (Actual)
Dates: Start 2001-10-16 (Actual); Primary Completion 2005-04-13 (Actual); Study Completion 2005-04-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of continued dosing with ALX1-11, up to a maximum of 24 months, in postmenopausal osteoporotic women who participated in Protocol ALX1-11-93001 (TOP). | 24 months of treatment

SECONDARY OUTCOMES:
To evaluate the continued efficacy of once-daily treatment with ALX1-11 for maintaining increases in BMD and other measures of bone quality and strength. | 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (132):
- United States (84):
  - 'The University of Alabama at Birmingham, Birmingham, Alabama
  - 'Rheumatology Associates of North Alabama, Huntsville, Alabama
  - 'Radiant Research - Phoenix North, Phoenix, Arizona
  - 'Osteoporosis Medical Center, Beverly Hills, California
  - 'East Bay Clinical Trial Center, Concord, California
  - 'Loma Linda Osteoporosis Research Center, Loma Linda, California
  - Foundation for Osteoporosis Research, Oakland, California
  - 'Desert Medical Advances, Palm Desert, California
  - 'VA Palo Alto Health Care System, Palo Alto, California
  - 'Boling Clinical Trials, Rancho Cucamonga, California
  - 'S.D. Arthritis & Osteoporosis Medical Clinic, San Diego, California
  - 'Radiant Research - San Diego, San Diego, California
  - 'San Francisco General Hospital, San Francisco, California
  - 'Longmont Medical Research Network, Longmont, Colorado
  - 'Northeast Clinical Research, LLC, Hamden, Connecticut
  - 'RASF - Clinical Research Center, Boca Raton, Florida
  - 'The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - 'Florida Wellcare Alliance, Inverness, Florida
  - 'Renstar Medical Group, Ocala, Florida
  - 'The Arthritis Center, Palm Harbor, Florida
  - 'The Centre for Arthritis and Rheumatic Diseases, South Miami, Florida
  - 'Radiant Research - Stuart & LakeWorth, Stuart, Florida
  - 'Palm Beach Research Center, West Palm Beach, Florida
  - 'Radiant Research, Honolulu, Hawaii
  - 'Intermountain Orthopaedics, Boise, Idaho
  - Rush-Prebyterian-St.Luke's Medical Center, Chicago, Illinois
  - 'The University of Chicago, Chicago, Illinois
  - 'University Hospital & Outpatient Center, Indianapolis, Indiana
  - 'Mercy Arthritis and Osteoporosis Center, Des Moines, Iowa
  - 'Wichita Clinic, Wichita, Kansas
  - 'Ochsner Clinic, New Orleans, Louisiana
  - 'Maine Center for Osteoporosis Research & Education, Bangor, Maine
  - 'Bethesda Health Research Center, Bethesda, Maryland
  - 'The Osteoporosis and Clinical Trials Center, Cumberland, Maryland
  - 'Arthritis & Osteoporosis Center of Maryland, Frederick, Maryland
  - 'The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - 'Brigham & Women's Hospital, Boston, Massachusetts
  - 'Michigan Bone & Mineral Clinic, Detroit, Michigan
  - 'Desoto Family Medical Center, Olive Branch, Mississippi
  - 'St. John's Medical Research Group, Springfield, Missouri
  - 'Arthritis, Osteoporosis Muscle Skeletal Disease Center, Concord, New Hampshire
  - 'Anderson and Collins Clinical Research Inc., South Plainfield, New Jersey
  - 'New Mexico Clinical Research and Osteoporosis Center, Albuquerque, New Mexico
  - 'Lovelace Scientific Resources, Albuquerque, New Mexico
  - 'College of Physicians and Surgeons, Columbia University, New York, New York
  - 'Rochester Clinical Research Inc., Rochester, New York
  - 'Stony Brook Clinical Research Trials Center, Stony Brook, New York
  - 'Physicians Clinical Research Services, White Plains, New York
  - 'Duke University Medical Center, Durham, North Carolina
  - 'Odyssey Research Services, Bismarck, North Dakota
  - Michael J. Lillestol, Fargo, North Dakota
  - 'Altru Health Systems / Altru Research Center, Grand Forks, North Dakota
  - 'Odyssey Research Services, Minot, North Dakota
  - 'Cleveland Clinic Foundation, Cleveland, Ohio
  - 'David R. Mandel M.D. Inc., Mayfield, Ohio
  - 'Oklahoma Center for Arthritis Therapy & Research, Inc., Tulsa, Oklahoma
  - 'Osteoporosis Center, Medford, Oregon
  - 'Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - 'Thomas Jefferson University, Philadelphia, Pennsylvania
  - 'University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - 'Clinical Research Center of Reading LLP, West Reading, Pennsylvania
  - 'Radiant Research, Wyomissing, Pennsylvania
  - 'Rhode Island Hospital, Providence, Rhode Island
  - 'Roger Williams Medical Center, Providence, Rhode Island
  - 'Radiant Research, Anderson, South Carolina
  - 'Columbia Arthritis Center, PA, Columbia, South Carolina
  - 'Radiant Research, Greer, South Carolina
  - 'Rapid City Medical Center, Rapid City, South Dakota
  - 'Averna Research Institute, Sioux Falls, South Dakota
  - 'Brown Clinic, Watertown, South Dakota
  - 'Clinsearch, Chattanooga, Tennessee
  - 'Radiant Research/Dallas, Dallas, Texas
  - 'Breco Research Inc., Houston, Texas
  - 'Diabetes Center of the Southwest, Midland, Texas
  - 'Diabetes & Glandular Disease Research Associates, P.A., San Antonio, Texas
  - 'Radiant Research San Antonio, San Antonio, Texas
  - 'Salt Lake Women's Center, Sandy City, Utah
  - 'Fletcher Allan Health Center, UHC Campus 1, Burlington, Vermont
  - 'Center for Arthritis and Diabetes, Newport News, Virginia
  - 'National Clinical Research, Inc., Richmond, Virginia
  - 'MCV Physicians Program for Osteoporosis, Richmond, Virginia
  - 'Osteoporosis Research Group, Seattle, Washington
  - 'University of Wisconsin Medical Foundation, Madison, Wisconsin
  - 'Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (4):
  - 'IDIM, Buenos Aires, BUE
  - 'Centro Médico T.I.E.M.P.O, Buenos Aires, BUE
  - 'Hospital Ramos Mejía, Buenos Aires, BUE
  - 'Centro de Osteopatias Medicas, Capital Federal, CBA
- Brazil (6):
  - 'Universidade Federal do Paraná, Curitiba, Paraná
  - 'Hospital Santa Casa de Misericórdia do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - 'Hospital do Servidor Público do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - 'Universidade Federal de São Paulo, São Paulo, São Paulo
  - 'Instituto de Saúde e Bem Estar da Mulher, São Paulo, São Paulo
  - 'Hospital Heliópolis, São Paulo, São Paulo
- Canada (21):
  - 'Heritage Medical Research Clinic, Calgary, Alberta
  - Osteoporosis Research Center, Vancouver, British Columbia
  - 'Manitoba Clinic, Winnipeg, Manitoba
  - Charlton medical Centre, Hamilton, Ontario
  - Rafat Faraawi, Kitchener, Ontario
  - 'Centre for Activity and Aging, London, Ontario
  - St. Joseph's Health Centre, London, Ontario
  - 'Royal Victoria Hospital, Montreal, Ontario
  - Oakville Bone Center, Oakville, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - 'Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - 'St. Michael's Hospital, Toronto, Ontario
  - 'Osteoporosis Research Program, Toronto, Ontario
  - Jude F. Rodrigues, Windsor, Ontario
  - 'Riverside Medical Centre, Charlottetown, Prince Edward Island
  - 'Complexe Hospitalier de la Sagami, Chicoutimi, Quebec
  - 'Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - 'Centre de Recherche du CHUM - Hopital Saint-Luc, Montreal, Quebec
  - Centre de recherche - CORQ, Sainte-Foy, Quebec
  - Novabyss Research Clinic, Sherbrooke, Quebec
  - 'Saskatoon Osteoporosis Centre, Saskatoon, Saskatchewan
- Israel (6):
  - 'Soroka Medical Center, Beersheba
  - 'Rambam Medical Center, Haifa
  - 'Lin Medical Center, Haifa
  - 'Hadassah University Hospital, Jerusalem
  - 'Chaim Sheba Medical Center, Ramat Gan
  - 'Lis Maternity Hospital, Tel Aviv
- Mexico (8):
  - 'Hospital Angeles de las Lomas, Huixquilucan, EMEX
  - 'Hospital Aranda de la Parra, León, Guanajuato
  - 'OPD Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara, Jalisco
  - 'Hospital Civil de Belem, Guadalajara, Jalisco
  - 'Medica Monraz, Guadalajara, Jalisco
  - 'Instituto Mexicano de Investigacion Clinica, Mexico City, Mexico City
  - 'Hospital de Mexico, Mexico City, Mexico City
  - 'Hospital Universitario de Monterrey, Monterrey Nuevo Leon
- 'Spitalul Clinic Judetean Cluj-Napoca, Cluj-Napoca, Romania
- Russia (2):
  - 'Scientific Center of Endocrinology of RAMS, Moscow
  - 'Russian Academy for Advanced Medical Studies, Moscow